CLINICAL TRIAL: NCT06046118
Title: Outcomes of Photobiomodulation in DRy Age Related macUlar Degeneration: a proSpective multicEnter raNdomized Controlled (DRUSEN) Study
Brief Title: Photobiomodulation in Dry Age Related Macular Degeneration
Acronym: DRUSEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Giuseppe Giannaccare, Professor, Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBM AMD
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age related Macular Degeneration; Photobiomodulation
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Two cycles of treatment using continuous and pulsed yellow light followed by continuous and pulsed red light.
  Cycle 1 consists of 8 sessions (two sessions per week for 4 weeks) and cycle 2 consists of 6 sessions (two sessions per week for 3 weeks).
  Interventions: Device: Yellow and red light emitting diode photobiomodulation (Eye Light, Espansione Group, Bologna, Italy)
- Sham group (Sham Comparator): Sham treatment will occur using a sham mask, designed to release a very low level of light, in this way the patient will not be able to distinguish if he is receiving the treatment or not.
  Cycle 1 consists of 8 sessions (two sessions per week for 4 weeks) and cycle 2 consists of 6 sessions (two sessions per week for 3 weeks).
  Interventions: Device: Sham Mask

INTERVENTIONS:
Device: Yellow and red light emitting diode photobiomodulation (Eye Light, Espansione Group, Bologna, Italy) — Each session consists of:
  * 1st phase: 300 seconds of continuous Yellow light (eyes closed) + 60 seconds of pulsed Yellow light (eyes opened)
  * 2nd phase: 300 seconds of continuous Red light(eyes closed) + 60 seconds of pulsed Red light (eyes opened).
  Cycle 1: 8 sessions (two PBM per week for 4 weeks); Cycle 2: 6 sessions (two PBM per week for 3 weeks).
  Arms: Treatment group
Device: Sham Mask — Low light emission mask (Sham Mask, Espansione group, Bologna, Italy)
  Arms: Sham group

SUMMARY:
The goal of this clinical trial is to evaluate effects of consecutive Yellow and Red Light Emitting Diode photobiomodulation in dry age-related macular degeneration (AMD). The main questions it aims to answer are:

* Is Yellow and Red Light Emitting Diode photobiomodulation effective in decreasing drusen volume in patients affected by dry AMD?
* Does Yellow and Red Light Emitting Diode photobiomodulation increase visual acuity and contrast sensitivity in patients affected by dry AMD? Participants will be randomly assigned to a treatment or a sham group.

Treatment consists in two cycles with two phases each:

* 1st phase: 300 seconds of continuous Yellow light with eyes closed + 60 seconds of pulsed Yellow light with eyes opened;
* 2d phase: 300 seconds of continuous Red light with eyes closed + 60 seconds of pulsed Red light with eyes opened.

Cycle 1 consists of 8 sessions (two PBM per week for 4 weeks) and cycle 2 consists of 6 sessions (two PBM per week for 3 weeks).

Researchers will compare patients in the treatment group to those in the sham group to evaluate differences in objective signs and subjective symptoms of dry AMD.

ELIGIBILITY:
Inclusion Criteria:

* BCVA ETDRS > 40 L ETDRS at 4 meters
* Diagnosis of DRY AMD AREDS grade 2-3
* Ability to communicate well with the investigator and able to understand and comply with the requirements of the study

Exclusion Criteria:

* Concomitant epilepsy
* Neurological diseases
* Psychiatric pathologies
* Herpes virus infections
* Dense cataract
* Pregnancy
* Other significant ocular and/or retinal diseases

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity variation | 1 month, 2 months and 4 months after each cycle
  ETDRS letters
Drusen Volume Variation | 1 month, 2 months and 4 months after each cycle
  Based on SD-OCT Heidelberg
Contrast sensitivity variation | 1 month, 2 months and 4 months after each cycle
  Based on Pelli Robson chart

CONTACTS AND LOCATIONS:
Locations (7):
- University of Paris, Paris, France
- Italy (3):
  - Università degli Studi di Ferrara, Ferrara
  - Università degli studi della Campania Luigi Vanvitelli, Napoli
  - Università di Torino, Torino
- Turkey (Türkiye) (2):
  - University of Ankara, Ankara
  - Koç University Hospital, Koç
- Earlam and Christopher, Taunton, United Kingdom

REFERENCES:
- [Derived] Borrelli E, Coco G, Pellegrini M, Mura M, Ciarmatori N, Scorcia V, Carnevali A, Lucisano A, Borselli M, Rossi C, Reibaldi M, Ricardi F, Vagge A, Nicolo M, Forte P, Cartabellotta A, Hasanreisoglu M, Kesim C, Demirel S, Yanik O, Bernabei F, Rothschild PR, Farrant S, Giannaccare G. Safety, Tolerability, and Short-Term Efficacy of Low-Level Light Therapy for Dry Age-Related Macular Degeneration. Ophthalmol Ther. 2024 Nov;13(11):2855-2868. doi: 10.1007/s40123-024-01030-w. Epub 2024 Sep 13. PMID 39271642